CLINICAL TRIAL: NCT01624506
Title: Observational Study of Anti-Reflux Surgery: Clinical Experience With the LINX Reflux Management System and Fundoplication
Brief Title: Observational Study of Anti-Reflux Surgery
Status: Completed | Type: Observational
Sponsor: Torax Medical Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 2776
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: GERD; Gastroesophageal Reflux; Gastro Esophageal Reflux
Keywords: Gastroesophageal Reflux Disease; Fundoplication; Magnetic Sphincter Augmentation; Proton Pump Inhibitors; GERD; PPI; MSA
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Magnetic Sphincter Augmentation: Patients will be treated with magnetic sphincter augmentation via the LINX Reflux Management System
- Fundoplication: Patients treated with laparoscopic fundoplication

SUMMARY:
The Anti-Reflux Surgical Study has been established to:

* Collect data about anti-reflux surgical treatment options (magnetic sphincter augmentation and Fundoplication) in everyday clinical practice
* Track the clinical course of patients from pre-operative assessment to three years post-surgery

DETAILED DESCRIPTION:
This study will track and monitor patients treated with either the magnetic sphincter augmentation or Fundoplication, making it the first Registry to collect data on both anti-reflux surgical options in the setting of everyday clinical experience.

ELIGIBILITY:
Inclusion Criteria:

* Individuals treated with LINX Reflux Management System or Fundoplication
* Individuals who have provided appropriate authorization per institutional policy and procedure to have clinical and health information collected for the Anti-Reflux Surgical Registry.
* Individuals willing to complete questionnaires and comply with the three years of follow-up.

Exclusion Criteria:

* Known circumstances that would make it unlikely for an individual to complete the three year follow-up (e.g. life expectancy <3 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing antireflux surgery for the treatment of gastroesophageal reflux disease (GERD)
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- Austria (2):
  - AKH Wien, Vienna
  - Herz Jesu Krankenhaus, Vienna
- Germany (13):
  - MIC Klinik Berlin, Berlin
  - Knappschafts Krankenhaus Bottrop, Bottrop
  - Diako Bremen, Bremen
  - Krankenhaus Castrop Rauxel, Castrop-Rauxel
  - Uniklinikum Koln, Cologne
  - Klinikum Forchheim, Forchheim
  - Krankenhaus Herne, Herne
  - Marien Krankenhaus, Kassel
  - Arabella Klinik, München
  - Ruppiner Kliniken, Neuruppin
  - Stadtkrankenhaus Schwabach, Schwabach
  - St. Rochus, Telgte
  - Ev. K Zweibrucken, Zweibrücken
- Policlinico San Donato, Milan, Italy
- United Kingdom (5):
  - Reflux Centre, Birmingham
  - Epsom and St. Helier Hospital, Epsom
  - Royal Devon & Exeter Hospital, Exeter
  - Spire Tunbridge Wells Hospital, Royal Tunbridge Wells
  - Weymouth Hospital, Weymouth

REFERENCES:
- [Derived] Bonavina L, Horbach T, Schoppmann SF, DeMarchi J. Three-year clinical experience with magnetic sphincter augmentation and laparoscopic fundoplication. Surg Endosc. 2021 Jul;35(7):3449-3458. doi: 10.1007/s00464-020-07792-1. Epub 2020 Jul 16. PMID 32676727
- [Derived] Riegler M, Schoppman SF, Bonavina L, Ashton D, Horbach T, Kemen M. Magnetic sphincter augmentation and fundoplication for GERD in clinical practice: one-year results of a multicenter, prospective observational study. Surg Endosc. 2015 May;29(5):1123-9. doi: 10.1007/s00464-014-3772-7. Epub 2014 Aug 30. PMID 25171881

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Not required
Period: Overall Study
Arm/Group | Magnetic Sphincter Augmentation | Fundoplication
Started | 530 | 230
Completed | 465 | 213
Not Completed | 65 | 17
Not completed — Lost to Follow-up | 29 | 15
Not completed — Withdrawal by Subject | 9 | 2
Not completed — Death | 1 | 0
Not completed — LINX explants | 23 | 0
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnetic Sphincter Augmentation | Fundoplication | Total
Number analyzed (Participants) | 530 | 230 | 760
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data not available for remaining subjects
  years
    number analyzed (Participants) | 517 | 210 | 727
    (all) | 46.8 (13.7) | 55.8 (12.1) | 49.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not available for remaining subjects
  Participants
    number analyzed (Participants) | 519 | 215 | 734
    Female | 198 | 113 | 311
    Male | 321 | 102 | 423
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 27 | 34 | 61
  Italy | 104 | 37 | 141
  United Kingdom | 101 | 26 | 127
  Germany | 298 | 133 | 431
Years with Gastroesophageal Reflux Disease (GERD) [Mean (Standard Deviation); unit: years] — Population: Data not available for remaining subjects
  years
    number analyzed (Participants) | 518 | 207 | 725
    (all) | 9.0 (7.9) | 8.9 (8.1) | 9.0 (7.9)
Years with Proton Pump Inhibitors (PPI) [Mean (Standard Deviation); unit: years] — Population: Data not collected for remaining subjects
  years
    number analyzed (Participants) | 517 | 203 | 720
    (all) | 6.1 (5.4) | 5.8 (5.7) | 6.0 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Gastroesophageal Reflux Disease Health Related Quality of Life Outcome (GERD-HRQL)
Description: Gastroesophageal Reflux Disease Health Related Quality of Life Outcomes (GERD-HRQL) Total scores range from 0-50 (min/max) 10 questions total, each rating 0-5 (min/max) Lower is better; higher is worse
Time Frame: 3 years post-surgery
Population: Enrolled subjects who completed the 3-year visit and responded to the Gastroesophageal Reflux Disease Health Related Quality of Life Outcome (GERD-HRQL) questionnaire are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Magnetic Sphincter Augmentation | Fundoplication
Number analyzed (Participants) | 328 | 97
score on a scale | 4.2 (5.7) | 4.9 (7.8)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Magnetic Sphincter Augmentation | Fundoplication
All-Cause Mortality (participants affected / at risk) | 1/530 | 0/230
Serious Adverse Events (participants affected / at risk) | 22/530 | 4/230
Other Adverse Events (participants affected / at risk) | 98/530 | 30/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnetic Sphincter Augmentation (N=530) | Fundoplication (N=230)
Device erosion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 10 (11) | 0 (0)
Gatric pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Worsening of GERD (Gastrointestinal disorders) | 6 (6) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnetic Sphincter Augmentation (N=530) | Fundoplication (N=230)
Heartburn (Gastrointestinal disorders) | 52 (61) | 14 (15)
Dysphagia (Gastrointestinal disorders) | 49 (54) | 16 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other